CLINICAL TRIAL: NCT05711485
Title: Clinical and Translational Investigations of Severe Malaria Pathophysiology [Parent Study Protocol]
Brief Title: Platelet-Directed Whole Blood Transfusion Strategy for Malaria
Acronym: PLATFORM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Johns Hopkins University (Other); Tropical Diseases Research Centre (Unknown); University of California, San Francisco (Other); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00015011
Record Dates: First submitted 2023-01-16; First posted 2023-02-03 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Severe Malaria; Thrombocytopenia
Keywords: Malaria; Plasmodium falciparum; Zambia
MeSH Terms: conditions — Malaria; Thrombocytopenia; Malaria, Falciparum | interventions — Exchange Transfusion, Whole Blood

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole blood transfusion (Experimental): Whole blood transfusion x1 (20 mL/kg)
  Interventions: Other: Whole blood transfusion
- Control (No Intervention): Standard-of-care

INTERVENTIONS:
Other: Whole blood transfusion — Whole blood is sourced from the Zambia National Blood Transfusion Service.
  Arms: Whole blood transfusion

SUMMARY:
Open-label randomized controlled trial to test the effectiveness of whole blood transfusion for improving survival in children with severe malaria complicated by thrombocytopenia.

DETAILED DESCRIPTION:
The PLATFORM trial is a single-center, open-label randomized controlled trial of whole blood transfusion for severe malaria complicated by thrombocytopenia. The trial will recruit 132 Zambian children 6 months to 15 years old with severe malaria defined according to modified WHO criteria with concomitant thrombocytopenia, defined here as a platelet count ≤75,000/uL, who do not otherwise have a current indication for transfusion according to current guidelines. Children will be randomized 1:1 to whole blood transfusion or no whole blood transfusion and followed to hospital discharge or death. The trial is nested within the Children and Adults with Severe Malaria (CHASM) cohort, a prospective observational study of severe malaria.

ELIGIBILITY:
Inclusion Criteria:

* Age <5 years
* Platelet count ≤75,000/uL
* Hemoglobin >5 and ≤9 g/dL
* P. falciparum parasitemia ≥500 parasites/uL
* Diagnosis of severe malaria meeting World Health Organization (WHO) criteria
* Ability and willingness of the legal guardian to comply with study protocol for the duration of the study
* Residence within health clinic catchment area
* Signed informed consent obtained from the parent or legal guardian of the participant

Exclusion Criteria:

* Residence in foster care or children otherwise under government supervision
* Residence outside the hospital catchment area, or plan to leave the area
* Presence of any other condition or abnormality which, in the opinion of the investigator, would compromise the safety of the participant or the quality of the data
* Any contraindication to whole blood transfusion

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2024-02-24 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of all-cause mortality | Up to hospital discharge or in-hospital death, up to 28 days on average
  Death due to any cause

SECONDARY OUTCOMES:
Change in hemoglobin (Hb) | Pre- and post-transfusion, comparing baseline measurements to measurements taken 2 hours after transfusion completion and 24 hours later. For the Control arm, measurements will be made at baseline and Study Hour 6 ±2 and 24 hours later
  The difference in Hb concentration between baseline (pre-transfusion) and post-transfusion
Change in platelet count | Pre- and post-transfusion, comparing baseline measurements to measurements taken 2 hours after transfusion completion and 24 hours later. For the Control arm, measurements will be made at baseline and Study Hour 6 ±2 and 24 hours later
  The difference in the platelet count between baseline (pre-transfusion) and post-transfusion
Change in white blood cell (WBC) count | Pre- and post-transfusion, comparing baseline measurements to measurements taken 2 hours after transfusion completion and 24 hours later. For the Control arm, measurements will be made at baseline and Study Hour 6 ±2 and 24 hours later
  The difference in the WBC count between baseline (pre-transfusion) and post-transfusion
Incidence of transfusion reaction | During or after transfusion, up to the day of hospital discharge or in-hospital death, up to 28 days on average
  Transfusion reactions (e.g., hypersensitivity, TACO, TRALI) graded on severity and likeliness of being related to transfusion
Length of hospitalization | Up to hospital discharge or in-hospital death, up to 28 days on average
  Interval in days from date of admission to date of discharge/death
Parasite clearance | 0-72 hours, measured every 12±2 hours
  Time to microscopic conversion to negative

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Ippolito, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States
- Tropical Diseases Research Centre, Ndola, Copperbelt, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to other researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Approx. 1-2 years after data collection

REFERENCES:
- [Background] Ippolito MM, Kabuya JB, Hauser M, Kamavu LK, Banda PM, Yanek LR, Malik R, Mulenga M, Bailey JA, Chongwe G, Louis TA, Shapiro TA, Moss WJ; Southern and Central Africa International Centers of Excellence for Malaria Research. Whole Blood Transfusion for Severe Malarial Anemia in a High Plasmodium falciparum Transmission Setting. Clin Infect Dis. 2022 Nov 30;75(11):1893-1902. doi: 10.1093/cid/ciac304. PMID 35439307